CLINICAL TRIAL: NCT02220842
Title: A Phase Ib Study of the Safety and Pharmacology of Atezolizumab Administered With Obinutuzumab in Patients With Relapsed/Refractory Follicular Lymphoma or Atezolizumab Administered With Obinutuzumab or Tazemetostat in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Safety and Pharmacology Study of Atezolizumab (MPDL3280A) Administered With Obinutuzumab or Tazemetostat in Participants With Relapsed/Refractory Follicular Lymphoma and Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29383; 2014-001812-21 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-20 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — atezolizumab; obinutuzumab; tazemetostat

ARMS (5):
- Arm 1 Cohort A (Safety Evaluation):Atezolizumab + Obinutuzumab (Experimental): Relapsed/refractory FL and DLBCL participants will receive obinutuzumab alone on Days 1, 8, and 15 of Cycle 1 (Cycle length = 21 days), followed by atezolizumab and obinutuzumab on Day 1 of Cycles 2-8, and then atezolizumab alone on Day 1 of Cycle 9 and every cycle thereafter until unacceptable toxicities or disease progression.
  Interventions: Drug: Atezolizumab; Drug: Obinutuzumab
- Arm 1 Cohort B (Expansion): Atezolizumab + Obinutuzumab (Experimental): Relapsed/refractory FL participants will receive atezolizumab and obinutuzumab as per schedule and dose decided from the safety evaluation stage, until unacceptable toxicities or disease progression.
  Interventions: Drug: Atezolizumab; Drug: Obinutuzumab
- Arm 1 Cohort C (Expansion): Atezolizumab + Obinutuzumab (Experimental): Relapsed/refractory DLBCL participants will receive atezolizumab and obinutuzumab as per schedule and dose decided from the safety evaluation stage, until unacceptable toxicities or disease progression.
  Interventions: Drug: Atezolizumab; Drug: Tazemetostat
- Arm 2 Cohort D (Safety Evaluation):Atezolizumab + Tazemetostat (Experimental): Relapsed/refractory DLBCL participants will receive atezolizumab (on Day 1) and tazemetostat (on Days 1-21) of each 21-day cycle until unacceptable toxicities or disease progression.
  Interventions: Drug: Atezolizumab; Drug: Tazemetostat
- Arm 2 Cohort E (Expansion): Atezolizumab + Tazemetostat (Experimental): Relapsed/refractory DLBCL participants will receive atezolizumab and tazemetostat as per schedule and dose decided from the safety evaluation stage, until unacceptable toxicities or disease progression.
  Interventions: Drug: Atezolizumab; Drug: Tazemetostat

INTERVENTIONS:
Drug: Atezolizumab — During safety evaluation stage, atezolizumab will be administered as 1200 milligrams (mg) intravenous (IV) infusion. During expansion stage, atezolizumab will be administered as either 1200 mg IV infusion or at dose decided from safety evaluation stage.
  Other Names: Tecentriq
Drug: Obinutuzumab — During safety evaluation stage, obinutuzumab will be administered as 1000 mg IV infusion. During expansion stage, obinutuzumab will be administered as either 1000 mg IV infusion or at dose decided from safety evaluation stage.
  Arms: Arm 1 Cohort A (Safety Evaluation):Atezolizumab + Obinutuzumab; Arm 1 Cohort B (Expansion): Atezolizumab + Obinutuzumab
Drug: Tazemetostat — Tazemetostat 800 mg will be administered orally, twice daily, on Days 1 to 21.
  Other Names: EPZ6438
  Arms: Arm 1 Cohort C (Expansion): Atezolizumab + Obinutuzumab; Arm 2 Cohort D (Safety Evaluation):Atezolizumab + Tazemetostat; Arm 2 Cohort E (Expansion): Atezolizumab + Tazemetostat

SUMMARY:
This open-label, multicenter, global study is designed to assess the safety, tolerability, preliminary efficacy, and pharmacokinetics of intravenous atezolizumab (MPDL3280A) and obinutuzumab in participants with refractory or relapsed follicular lymphoma (FL) or atezolizumab and obinutuzumab or tazemetostat administered in participants with refractory or relapsed diffuse large B-cell lymphoma (DLBCL). The anticipated duration of this study is approximately 4.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, CD20-positive, relapsed or refractory (defined as having relapsed within 6 months to the previous treatment) FL or DLBCL (including primary mediastinal large B-cell lymphoma [PMLBCL])
* Bone marrow biopsy at screening (unless it was performed within 3 months prior to screening)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Life expectancy greater than or equal to (>=) 12 weeks
* Has a QT interval corrected by Fridericia's formula (QTcF) less than or equal to (<=) 480 milliseconds (msec)
* At least one bi-dimensionally measurable nodal lesion >1.5 cm in its longest diameter by computed tomography (CT) scan or MRI, as defined by the Lugano Classification
* Adequate hematologic and end-organ function
* Archival tumor tissue
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of atezolizumab or 18 months after the last dose of obinutuzumab, whichever is longer
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

* Known central nervous system lymphoma, leptomeningeal lymphoma, or histologic evidence of transformation from an indolent lymphoma to a high-grade or DLBCL
* Grade 3b FL, small lymphocytic lymphoma (SLL), or Waldenström's macroglobulinemia (WM) or other lymphoma subtypes except as stated in the inclusion criteria
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently); participants with indwelling catheters are eligible
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Has had prior exposure to tazemetostat or other inhibitor(s) of enhancer of zeste homolog 2 (EZH2)
* Regular treatment with corticosteroids within the 2 or 4 weeks prior to the start of Cycle 1, unless administered for indications other than non-Hodgkin's lymphoma at a dose equivalent to < 30 mg/day prednisone/prednisolone
* Pregnant and lactating women
* History of autoimmune disease
* Participants with history of confirmed progressive multifocal leukoencephalopathy (PML)
* Participants with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest CT scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed
* Positive test for Human Immunodeficiency Virus (HIV)
* History of chronic hepatitis B infection or positive test results for active or chronic hepatitis B or hepatitis C
* Significant cardiovascular disease, such as cardiac disease (New York Heart Association Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina
* Hypersensitivity or prior treatment with obinutuzumab
* Fludarabine or Campath within 12 months prior to study entry
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including but not limited to interferon, interleukin-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1
* Treatment with systemic immunosuppressive medications, including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents within 2 weeks prior to Cycle 1, Day 1; inhaled corticosteroids and mineralocorticoids are allowed
* Participants with active tuberculosis (TB) will be excluded from the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities (DLTs) | 21 days (for Arm 1: Days 1 to 21 to Cycle 2; for Arm 2: Days 1 to 21 of Cycle 1, cycle length = 21 days)
Recommended Phase 2 Dose (RP2D) of Atezolizumab | 21 days (for Arm 1: Days 1 to 21 to Cycle 2; for Arm 2: Days 1 to 21 of Cycle 1, cycle length = 21 days)

SECONDARY OUTCOMES:
Obinutuzumab Minimum Serum Concentration (Cmin) | Preinfusion (hour 0) on Day 1, 8, 15 of Cycle 1, Day 1 of Cycles 2, 3, 4, 6, 8, every 8 cycles thereafter up to treatment discontinuation, 120 days after treatment discontinuation (treatment discontinuation=up to approx 57 weeks) (Cycle=21 days)
Percentage of Participants With Adverse Events (AEs) Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) | Baseline up to approximately 4.5 years
Percentage of Participants With Anti-therapeutic Antibody Response to Atezolizumab and Obinutuzumab | Baseline up to approximately 4.5 years
Atezolizumab Maximum Serum Concentration (Cmax) | Preinfusion (hour 0) on Day 1 of Cycle 1 up to approx 57 weeks (detailed timeframe is provided in outcome description section)
  Arm 1: preinfusion (hour 0) on Day 1 of Cycle 1, 30 minutes post end of atezolizumab infusion (infusion over 30-60 minutes) on Day 1 of Cycle 2, preinfusion on Day 1 of Cycles 3, 4, 6, 8, and every 8 cycles thereafter up to treatment discontinuation, 120 days after treatment discontinuation (treatment discontinuation=up to approx 57 weeks), additionally preinfusion on Day 1 of Cycle 9; Arm 2: preinfusion (hour 0) and 30 minutes post end of atezolizumab infusion (infusion over 30-60 minutes) on Day 1 of Cycles 1 and 3, preinfusion on Day 1 of Cycles 2, 8, every 8 cycles thereafter up to treatment discontinuation, 120 days after treatment discontinuation (treatment discontinuation=up to approx 57 weeks) (Cycle=21 days)
Atezolizumab Minimum Serum Concentration (Cmin) | Preinfusion (hour 0) on Day 1 of Cycle 1 up to approx 57 weeks (detailed timeframe is provided in outcome description section)
  Arm 1: preinfusion (hour 0) on Day 1 of Cycles 1, 3, 4, 6, 8, and every 8 cycles thereafter up to treatment discontinuation, 120 days after treatment discontinuation (treatment discontinuation=up to approx 57 weeks), pre-infusion on Day 1 of Cycle 9; Arm 2: preinfusion (hour 0) on Day 1 of Cycles 1, 2, 3, 8, every 8 cycles thereafter up to treatment discontinuation, 120 days after treatment discontinuation (treatment discontinuation=up to approx 57 weeks) (Cycle = 21 days)
Obinutuzumab Maximum Serum Concentration (Cmax) | Arm 1: Preinfusion (hour 0) on Day 1 of Cycle 1 up to approx 57 weeks (detailed timeframe is provided in outcome description section)
  Arm 1: preinfusion (hour 0) on Day 1, 4-hour post start of infusion on Day 2, preinfusion (hour 0) and 4-hour post start of infusion on Day 8, 15 of Cycle 1, Day 1 of Cycles 2, 3, 4, 6, 8, every 8 cycles thereafter up to treatment discontinuation, 120 days after treatment discontinuation (treatment discontinuation=up to approx 57 weeks) (Cycle=21 days)
Percentage of Participants With Best Overall Response According to Lugano Classification | Cycle 3 Day 15 (Cycle 4 Day 15 for Arm 1) up to progression of disease, death, or withdrawal of consent, whichever occurs first (up to approximately 4.5 years) (Cycle=21 days)
Percentage of Participants With Objective Response (Complete Response or Partial Response) According to Lugano Classification | Cycle 3 Day 15 (Cycle 4 Day 15 for Arm 1) up to progression of disease, death, or withdrawal of consent, whichever occurs first (up to approximately 4.5 years) (Cycle=21 days)
Progression Free Survival (PFS) According to Lugano Classification | Cycle 3 Day 15 (Cycle 4 Day 15 for Arm 1) up to progression of disease, death, or withdrawal of consent, whichever occurs first (up to approximately 4.5 years) (Cycle=21 days)
Overall Survival (OS) | Baseline until death due to any cause (up to approximately 4.5 years)
Duration of Objective Response (DOR) According to Lugano Classification | From first documented complete or partial response up to progression of disease, death, or withdrawal of consent, whichever occurs first (up to approximately 4.5 years)
Tazemetostat Plasma Concentrations | Arm 2: predose (hour 0) on Day 1 of Cycles 1, 2, 3, 4, 8, every 8 cycles thereafter up to Cycle 17; 1, 2, 4 hours post dose on Day 1 of Cycles 1 and 3; additionally (in Cohort E only) 0.5, 6, 8 hours post dose on Cycle 3 Day 1 (Cycle=21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - UW- Fred Hutchinson Cancer Center, Seattle, Washington
- France (5):
  - Hopital Claude Huriez - CHU Lille; Service des maladies du sang, Lille
  - Hopital Saint Eloi, Montpellier
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany
- Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont, Italy
- Barts Hospital, London, United Kingdom

REFERENCES:
- [Derived] Palomba ML, Cartron G, Popplewell L, Ribrag V, Westin J, Huw LY, Agarwal S, Shivhare M, Hong WJ, Raval A, Chang AC, Penuel E, Morschhauser F. Combination of Atezolizumab and Tazemetostat in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma: Results From a Phase Ib Study. Clin Lymphoma Myeloma Leuk. 2022 Jul;22(7):504-512. doi: 10.1016/j.clml.2021.12.014. Epub 2021 Dec 24. PMID 35151584
- [Derived] Palomba ML, Till BG, Park SI, Morschhauser F, Cartron G, Marks R, Shivhare M, Hong WJ, Raval A, Chang AC, Penuel E, Popplewell LL. Combination of Atezolizumab and Obinutuzumab in Patients with Relapsed/Refractory Follicular Lymphoma and Diffuse Large B-Cell Lymphoma: Results from a Phase 1b Study. Clin Lymphoma Myeloma Leuk. 2022 Jul;22(7):e443-e451. doi: 10.1016/j.clml.2021.12.010. Epub 2021 Dec 24. PMID 35031227